CLINICAL TRIAL: NCT00625391
Title: GTP and Tai Chi for Bone Health: a Pilot Study
Brief Title: Green Tea and Tai Chi for Bone Health
Acronym: GTP-TC-Bone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Leslie Shen, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R21AT003735-01A1 (NIH); R21AT003735-01A1 (NIH)
Record Dates: First submitted 2008-02-26; First posted 2008-02-28 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Osteoporosis
Keywords: postmenopausal, bone, dietary supplement, mind-body exercise
MeSH Terms: conditions — Osteoporosis | interventions — Tea; rac1 GTP-Binding Protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo pill (Placebo Comparator): 24 weeks of placebo.
  Interventions: Drug: Placebo
- Green Tea Polyphenols (GTP) (Active Comparator): 24 weeks of green tea polyphenols
  Interventions: Drug: Green Tea Polyphenols (GTP)
- Placebo+Tai Chi (TC) (Active Comparator): 24 weeks of placebo plus Tai Chi exercise.
  Interventions: Drug: Placebo+Tai Chi (TC)
- GTP+TC (Active Comparator): 24 weeks of green tea polyphenols plus Tai Chi exercise.
  Interventions: Drug: GTP+TC

INTERVENTIONS:
Drug: Placebo — 500 mg medicinal starch pills daily
  Other Names: Placebo control group
  Arms: Placebo pill
Drug: Green Tea Polyphenols (GTP) — 500 mg green tea polyphenols daily
  Other Names: Green tea polyphenols group
  Arms: Green Tea Polyphenols (GTP)
Drug: Placebo+Tai Chi (TC) — 500 mg medicinal starch daily and Tai Chi (3x/week) for 24 weeks
  Other Names: Placebo plus tai chi exercise group
  Arms: Placebo+Tai Chi (TC)
Drug: GTP+TC — 500 mg GTP daily plus TC exercise (3x/week) for 24 weeks
  Other Names: Green tea polyphenols plus tai chi exercise group
  Arms: GTP+TC

SUMMARY:
Osteoporosis is a major health problem in postmenopausal women. Our long-term goal is to develop a new alternative treatment that include a dietary supplement (green tea extract) and a mind-body exercise (Tai Chi) for lessening bone loss in postmenopausal women with low bone mass. A combination of dietary supplement and moderate intensity exercise now becomes a new alternative treatment in reducing bone loss in postmenopausal women with low bone mass, due to the possible stronger effects of the combination than individual treatments. Objective: To test a CAM intervention including green tea polyphenol (GTP) and Tai Chi (TC) exercise for feasibility, and to quantitatively assess their individual and conjugate effects on postmenopausal women with osteopenia. Hypotheses: (1) 24 weeks of GTP supplement, TC exercise, and their combination will benefit bone remodeling as measured by bone biomarkers and muscle strength/physical function in postmenopausal women with osteopenia compared to those receiving placebo only, and (2) the changes in bone biomarkers associated with bone remodeling will be correlated with the changes in oxidative stress.

DETAILED DESCRIPTION:
This is a 24-week, randomized, and placebo-controlled intervention trial to investigate the effects of green tea polyphenols (GTP) and Tai Chi (TC) on relevant primary and secondary endpoints in postmenopausal women with osteopenia. Women at least 2 years after menopause, with osteopenia, will be recruited primarily from local senior independent/assisted living facilities, municipal senior community centers, and obstetrics and gynecology clinics. After screening, qualified participants will be matched for age and will be randomly assigned to one of the four treatment groups: placebo, GTP, placebo+TC, and GTP+TC. During the 24-week intervention, all participants will be provided with calcium and vitamin D daily. The participants in the placebo group will receive medicinal starch for 24 weeks. The GTP participants will receive GTP for 24 weeks. The placebo+TC participants will receive both placebo and TC treatments for 24 weeks. The GTP+TC participants will receive both GTP and TC treatments for 24 weeks. Participants will receive the primary and secondary outcome measures at baseline, 4, 12, and 24 weeks. The primary outcome measures are concentrations of bone biomarkers. The secondary outcome measure is a biomarker of oxidative stress DNA damage. Additional secondary outcome is muscle strength/physical function. Investigators evaluating the endpoints will be blinded to intervention allocation.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 2 years after menopause (to ensure established postmenopausal status).
* Sedentary at baseline.
* Normal laboratory evaluation, thyroid function, hepatic function, renal function.
* Osteopenia.

Exclusion Criteria:

* History of scoliosis, severe osteoarthritis, etc., or other spinal disease that may result in anatomy unsuitable for accurate bone densitometry.
* History of cancer with some exceptions.
* History of metabolic bone disease.
* Having used anabolic steroids, calcitonin, calcitriol, alfacalcidol, etc.
* Fluoride treatment at a dose greater than 1 mg/day any time.
* History of glucocorticoid treatment.
* Any previous treatment with bisphosphonates.
* Uncontrolled intercurrent illness such as symptomatic congestive heart failure, myocardial infarction or stroke, hypertension, or terminal illness.
* Physical conditions that preclude participation of exercise intervention.
* Cognitive impairment.
* Depression.
* History of malabsorption syndrome and uncontrolled diabetes mellitus.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li (Leslie) Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Shen CL, Chyu MC, Yeh JK, Felton CK, Xu KT, Pence BC, Wang JS. Green tea polyphenols and Tai Chi for bone health: designing a placebo-controlled randomized trial. BMC Musculoskelet Disord. 2009 Sep 4;10:110. doi: 10.1186/1471-2474-10-110. PMID 19732445
- [Background] Shen CL, Yeh JK, Cao JJ, Chyu MC, Wang JS. Green tea and bone health: Evidence from laboratory studies. Pharmacol Res. 2011 Aug;64(2):155-61. doi: 10.1016/j.phrs.2011.03.012. Epub 2011 Apr 5. PMID 21473914
- [Background] Shen CL, Yeh JK, Cao JJ, Wang JS. Green tea and bone metabolism. Nutr Res. 2009 Jul;29(7):437-56. doi: 10.1016/j.nutres.2009.06.008. PMID 19700031
- [Background] Shen CL, Chyu MC, Wang JS. Tea and bone health: steps forward in translational nutrition. Am J Clin Nutr. 2013 Dec;98(6 Suppl):1694S-1699S. doi: 10.3945/ajcn.113.058255. Epub 2013 Oct 30. PMID 24172296
- [Result] Shen CL, Chyu MC, Yeh JK, Zhang Y, Pence BC, Felton CK, Brismee JM, Arjmandi BH, Doctolero S, Wang JS. Effect of green tea and Tai Chi on bone health in postmenopausal osteopenic women: a 6-month randomized placebo-controlled trial. Osteoporos Int. 2012 May;23(5):1541-52. doi: 10.1007/s00198-011-1731-x. Epub 2011 Jul 16. PMID 21766228
- [Result] Shen CL, Chyu MC, Pence BC, Yeh JK, Zhang Y, Felton CK, Doctolero S, Wang JS. Green tea polyphenols supplementation and Tai Chi exercise for postmenopausal osteopenic women: safety and quality of life report. BMC Complement Altern Med. 2010 Dec 9;10:76. doi: 10.1186/1472-6882-10-76. PMID 21143878
- [Result] Qian G, Xue K, Tang L, Wang F, Song X, Chyu MC, Pence BC, Shen CL, Wang JS. Mitigation of oxidative damage by green tea polyphenols and Tai Chi exercise in postmenopausal women with osteopenia. PLoS One. 2012;7(10):e48090. doi: 10.1371/journal.pone.0048090. Epub 2012 Oct 31. PMID 23118932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 2008 - December 2008. Location: community setting
Pre-assignment Details: There was no any significant events arranged.
Groups:
- Placebo Group: Placebo group receiving 500 mg medicinal starch daily for 24 weeks.
- Green Tea Polyphenols (GTP) Group: Green tea polyphenols (GTP) group receiving 500 mg of GTP per day for 24 weeks.
- Placebo + Tai Chi Group: Placebo+Tai Chi group receiving both placebo treatment and Tai Chi training (60-minute group exercise, 3 times per week)for 24 weeks.
- GTP + Tai Chi Group: GTP+Tai Chi group receiving both GTP and Tai Chi training for 24 weeks.
Period: Overall Study
Arm/Group | Placebo Group | Green Tea Polyphenols (GTP) Group | Placebo + Tai Chi Group | GTP + Tai Chi Group
Started | 44 | 47 | 42 | 38
Completed | 37 | 39 | 37 | 37
Not Completed | 7 | 8 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo group receiving 500 mg medicinal starch daily for 24 weeks.
- Green Tea Polyphenols (GTP): Green tea polyphenols (GTP) group receiving 500 mg of GTP per day for 24 weeks.
- Placebo+Tai Chi: Placebo+Tai Chi group receiving both placebo treatment and Tai Chi training (60-minute group exercise, 3 times per week)for 24 weeks.
- GTP+Tai Chi: GTP+Tai Chi group receiving both GTP and Tai Chi training for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Green Tea Polyphenols (GTP) | Placebo+Tai Chi | GTP+Tai Chi | Total
Number analyzed (Participants) | 44 | 47 | 42 | 38 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 42 | 36 | 33 | 149
  >=65 years | 6 | 5 | 6 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (7.5) | 56.5 (5.5) | 58.3 (7.7) | 57.6 (6.7) | 57.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 42 | 38 | 171
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 47 | 42 | 38 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (100%) in Ratio of Bone Formation Marker to Bone Resorption Marker
Description: Bone formation biomarker: bone-specific alkaline phosphatase (BAP) Bone resorption biomarker: tartrate-resistant acid phosphatase (TRAP)
Time Frame: 24 weeks
Population: Analyzed on those who completed the study. Percent change relative to the baseline for each group.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Placebo: Placebo group receiving 500 mg medicinal starch daily for 24 weeks.
  Green tea polyphenols (GTP) group receiving 500 mg of GTP per day for 24 weeks.
  placebo+Tai Chi group receiving both placebo treatment and Tai Chi training (60-minute group exercise, 3 times per week)for 24 weeks.
  GTP+Tai Chi group receiving both GTP and Tai Chi training for 24 weeks.
- Green Tea Polyphenols: GTP group receiving 500 mg green tea polyphenols daily for 24 weeks
- Placebo + Tai Chi: Placebo + Tai Chi: receiving 500 mg medicinal starch daily and group Tai Chi exercise (60 min/session, 3 sessions/week) for 24 weeks
- Green Tea Polyphenol + Tai Chi: GTP + Tai Chi: receiving 500 mg green tea polyphenols daily and group Tai Chi exercise (60 min/session, 3 sessions/week) for 24 weeks.
Arm/Group | Placebo | Green Tea Polyphenols | Placebo + Tai Chi | Green Tea Polyphenol + Tai Chi
Number analyzed (Participants) | 37 | 39 | 37 | 37
percentage change from baseline | 106.1 (3.7) | 103.6 (2.9) | 112.3 (3.0) | 113.0 (3.0)

2. Secondary Outcome: Oxidative Stress Damage Biomarker
Description: Oxidative stress damage biomarker: urinary 8-hydroxy-2'-deoxyguanosine (8-OHdG) test
Time Frame: 24 weeks
Population: Analyzed who completed the study.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Placebo | Green Tea Polyphenols | Placebo + Tai Chi | Green Tea Polyphenol + Tai Chi
Number analyzed (Participants) | 37 | 39 | 37 | 37
ng/mg creatinine | 73.5 (50.9) | 33.5 (33.1) | 29.7 (21.9) | 20.6 (19.8)

ADVERSE EVENTS:
Time Frame: 24 weeks during the study period.
Description: Total number of participants at risk "serious and other [Non-serious] adverse events.
Groups:
- Placebo: Medicinal starch at 500 mg daily for 24 weeks
- Green Tea Polyphenols (GTP): Green tea polyphenols at 500 mg daily for 24 weeks
- Placebo+Tai Chi (TC): Medicinal starch at 500 mg daily and Tai Chi group exercise at 1 hour/session x 3 sessions/week for 24 weeks
- GTP+TC: Green tea polyphenols at 500 mg daily and Tai Chi group exercise at 1 hour/session x 3 sessions/week for 24 weeks
Arm/Group | Placebo | Green Tea Polyphenols (GTP) | Placebo+Tai Chi (TC) | GTP+TC
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/39 | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
Limitation of this study included: (1) the number of subjects in each group at the baseline was not equal. (2) The amount of dietary calcium intake for each subject was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No